CLINICAL TRIAL: NCT07199257
Title: A Multicenter Clinical Trial Evaluating the Efficacy, Safety, Pharmacokinetics, and Immunogenicity of GR1802 Injection in Combination With Background Therapy in Patients With Seasonal Allergic Rhinitis.
Brief Title: A Study of GR1802 Injection in Patients With Seasonal Allergic Rhinitis.
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Genrix (Shanghai) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GR1802-015
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Allergic Rhinitis, Seasonal
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part one subjects received open-label treatment. Part two subjects received double-blind treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interleukin-4 receptor responder(Part One) (Experimental): Part one
  Interventions: Biological: GR1802 injection
- Interleukin-4 receptor responder(Part Two) (Experimental): Part two
  Interventions: Biological: GR1802 injection
- Placebo (Placebo Comparator): Part two
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: GR1802 injection — Recombinant fully human anti-IL4Rα monoclonal antibody drug.
  Arms: Interleukin-4 receptor responder(Part One); Interleukin-4 receptor responder(Part Two)
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Allergic rhinitis (AR) is a non-infectious chronic inflammatory disease of the nasal mucosa mainly mediated by immunoglobulin E after exposure to allergens in atopic individuals. The typical symptoms of AR are paroxysmal sneezing, watery rhinorrhea, itching, and nasal congestion, which may be accompanied by ocular symptoms, including eye itching, tearing, redness, and burning sensation, which are more common in patients with hay fever allergies.

ELIGIBILITY:
Main Inclusion Criteria:

1. Voluntarily sign the informed consent form.
2. Seasonal allergic rhinitis has been prevalent for at least 2 years.Positive for allergens associated with seasonal allergic rhinitis.
3. Poor control of seasonal allergic rhinitis with nasal glucocorticoids or other therapeutic agents during the same pollen season in the past.
4. Weight≥30kg.
5. Symptom severity scores for the season met the enrollment criteria.

Main Exclusion Criteria:

1. Other nasal comorbidities or co-morbidities/states that may be present at the time of screening that affect efficacy determination.
2. Subjects whose allergen exposures in their home or work environments may be expected to change significantly during the trial period.
3. Subjects with poorly controlled recent asthma conditions.
4. Presence of current or past history of infection of special concern, e.g., active tuberculosis, helminthic infections, severe herpes virus infections, etc.
5. Previous use of anti-interleukin 4 receptor alpha subunit (IL4Rα) monoclonal antibody.
6. Have a serious underlying medical condition that, in the opinion of the investigator, may pose a risk to subject safety by participation in a clinical trial.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs)(Part One) | up to 12 weeks
Change from Baseline in rTNSS( reflective total nasal symptom scores)(Part Two) | up to 2 weeks
  Scores range from 0 to 12, with higher scores indicating more severe symptoms.

SECONDARY OUTCOMES:
Change from Baseline in rTOSS( reflective total ocular symptom scores)(Part One/Two) | up to 2、4 weeks
  Scores range from 0 to 9, with higher scores indicating more severe symptoms.
Percentage Change from Baseline in rTNSS(Part One/Two) | up to 2、4 weeks
  Scores range from 0 to 12, with higher scores indicating more severe symptoms.
Mean change from baseline in iTNSS(instantaneous total nasal symptom scores)(Part One/Two) | week 2、4
  Scores range from 0 to 12, with higher scores indicating more severe symptoms.
Mean change from baseline in iTOSS(instantaneous total ocular symptom scores)(Part One/Two) | week 2、4
  Scores range from 0 to 9, with higher scores indicating more severe symptoms.
Change from baseline in RQLQ(Rhinoconjunctivitis Quality of Life Questionnaire) scores(Part One/Two) | week2、4
  There are 28 questions in 7 fields，Each question is answered on a 7-point scale (0 to 6).
Incidence of ADAs(Part One/Two) | up to 12 weeks
drug concentration、Ctrough(Part One/Two) | up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan university, Wuhan, Hubei, China